CLINICAL TRIAL: NCT02562391
Title: Effect of Left Atrial Appendage Excision on Procedure Outcome in Patients With Persistent and Long-standing Persistent Atrial Fibrillation Undergoing Surgical Ablation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9872TLAA
Record Dates: First submitted 2015-09-24; First posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; ablation; thoracoscopy; left atrial appendage
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PVI+Box lesions (Active Comparator): Patients were treated with video-assisted thoracoscopy under general anesthesia, according to a previously described protocol. In brief, PVI was performed from the epicardial side with a bipolar radiofrequency ablation clamp. At least 2 overlapping applications around each of the ipsilateral veins were made, and isolation was confirmed by the absence of PV potentials and exit block during pacing. In addition to PVI, the bilateral epicardial ganglia were found by high-frequency stimulation and ablated, as confirmed by the absence of a vagal response after ablation. Finally additional lines were made to create a posterior box lesion. Sensing and pacing maneuvers verified isolation of the posterior box.
  Interventions: Device: Surgical ablation of the left atrium (PVI+Box lesions)
- PVI+Box lesions+LAA cutting (Experimental): Patients were treated with video-assisted thoracoscopy under general anesthesia, according to a previously described protocol. In brief, PVI was performed from the epicardial side with a bipolar radiofrequency ablation clamp. At least 2 overlapping applications around each of the ipsilateral veins were made, and isolation was confirmed by the absence of PV potentials and exit block during pacing. In addition to PVI, the bilateral epicardial ganglia were found by high-frequency stimulation and ablated, as confirmed by the absence of a vagal response after ablation. Finally additional lines were made to create a posterior box lesion. Sensing and pacing maneuvers verified isolation of the posterior box.The left atrial appendage was removed by stapling and then cutting.
  Interventions: Device: Surgical ablation of the left atrium (PVI+Box lesions) and left atrial appendage cutting

INTERVENTIONS:
Device: Surgical ablation of the left atrium (PVI+Box lesions)
  Arms: PVI+Box lesions
Device: Surgical ablation of the left atrium (PVI+Box lesions) and left atrial appendage cutting
  Arms: PVI+Box lesions+LAA cutting

SUMMARY:
The aim of this study is to assess the effect of left atrial appendage excision on atrial fibrillation recurrence and incidence of stroke in patients with persistent and long-standing persistent atrial fibrillation undergoing surgical ablation.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with persistent and long-standing persistent atrial fibrillation eligible for thoracoscopy surgical ablation
* Signed inform consent

Key Exclusion Criteria:

* Paroxysmal atrial fibrillation
* Contraindications for surgical ablation
* Unwilling to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2011-05; Primary Completion 2015-05 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation recurrences | 18 months

CONTACTS AND LOCATIONS:
Locations (4):
- Russia (4):
  - Federal Center of Cardiovascular surgery, Krasnoyarsk
  - Federal State Institution Clinical Hospital of the Presidental Administration of the RF, Moscow
  - Scientific center of the cardiovascular surgery named by A.N. Bakulev, Moscow
  - State Research Institute of CIrculation Pathology, Novosibirsk

REFERENCES:
- [Derived] Romanov A, Pokushalov E, Elesin D, Bogachev-Prokophiev A, Ponomarev D, Losik D, Bayramova S, Strelnikov A, Shabanov V, Pidanov O, Kropotkin E, Ivanickii E, Karaskov A, Steinberg JS. Effect of left atrial appendage excision on procedure outcome in patients with persistent atrial fibrillation undergoing surgical ablation. Heart Rhythm. 2016 Sep;13(9):1803-9. doi: 10.1016/j.hrthm.2016.05.012. Epub 2016 May 12. PMID 27180620